CLINICAL TRIAL: NCT05685381
Title: Contextualizing Asthma Self-Management With Measures of Indoor Air Quality for Black Adults With Uncontrolled Asthma
Brief Title: Indoor Air Quality for Black Adults With Uncontrolled Asthma
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Maureen George, Professor of Nursing at the Columbia University Irving Medical Center, Columbia University
Other Study IDs: AAAT0939 - sub-study; 3R01NR019275-02S1 (NIH)
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Asthma
Keywords: Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases; Respiratory Hypersensitivity; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases; Greenhouse Effect; Air Pollution, Indoor
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases; Respiratory Hypersensitivity; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Black adults with persistent asthma in homes with gas kitchen appliances: Black adults with persistent asthma that reside in homes with kitchen appliances (i.e., cooktops, ovens, and ranges) fueled by combustible gas.
- Black adults with persistent asthma in homes without gas kitchen appliances: Black adults with persistent asthma that reside in homes with kitchen appliances (i.e., cooktops, ovens, and ranges) not fueled by combustible gas.

SUMMARY:
The aims of this project are twofold:

1. to characterize indoor air quality components obtained from apartments with gas stoves and open kitchens in a cohort of Black adults with uncontrolled asthma recruited from federally qualified health centers and enrolled in the parent study.
2. to conduct a comprehensive assessment of feasibility, implementation, and acceptability of the study.

DETAILED DESCRIPTION:
People spend as much as 90% of their time indoors, making indoor air quality (IAQ) particularly important to health. Many homes in New York City, particularly low-income housing, contain gas kitchen appliances, which generate fuel through the combustion of natural gas, generating indoor pollutants. Increasing evidence finds that even low levels of these pollutants are hazardous for human health. Those most vulnerable to ambient air pollution live in homes with gas appliances and inadequate ventilation. Moreover, individuals with pre-existing diseases like asthma are particularly susceptible to adverse health effects from poor IAQ, which gas stoves may exacerbate. This study addresses the important problem of uncontrolled asthma among a group at high risk for asthma and its adverse effects - Black adults who reside in homes with gas stoves and open kitchens. The investigator aims to characterize indoor air quality components in a cohort enrolled in the parent R01 (NCT05341726) and conduct a comprehensive assessment of feasibility including process, implementation and acceptability metrics. Identifying new targets for asthma self-management that could produce better health outcomes, thus addressing an important health inequity issue.

ELIGIBILITY:
Inclusion Criteria (participants):

Patient participants will

1. be adults (> or = 18 years of age)
2. self-report race as 'Black' race (African American, African, Caribbean, West Indian, multi-racial [Black AND one or more additional races]); identify their ethnicity as Hispanic OR non-Hispanic
3. have clinician-diagnosed persistent asthma (defined as being prescribed inhaled corticosteroids in the last 48 months) or have had an asthma exacerbation (e.g., ER visit, course of Prednisone) regardless of controller medicine use
4. receive asthma care at a partner federally qualified health center and
5. screen positive for uncontrolled asthma as measured by the Asthma Control Questionnaire- 6 items (ACQ-6) and erroneous beliefs as measured by the Conventional and Alternative Management for Asthma (CAM-A) survey.

Exclusion Criteria (participants):

1. non-English speaking or
2. serious mental health conditions that preclude completion of study procedures or confound analyses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Black adults with persistent asthma that receive care at partner federally qualified health centers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Completion of acceptability questionnaire | Post-trial visit (up to 3 months after intervention completion)
  The number of participants who complete the acceptability questionnaire. The acceptability questionnaire is a semi-structured interview at the time of indoor air quality sample retrieval and will be guided by the constructs of the Theoretical Framework of Acceptability (e.g., burden, user experience, attitudes, participation intentions).

CONTACTS AND LOCATIONS:
Overall Officials: Maureen George, PhD, Principal Investigator — Columbia University School of Nursing
Locations (2):
- United States (2):
  - Sun River Health, Beacon, New York
  - Bedford Stuyvesant Family Health Center, Brooklyn, New York

IPD SHARING:
Plan to Share IPD: No